CLINICAL TRIAL: NCT03734874
Title: Evaluation of the Effects of Hesperidin Supplementation in Patients With Metabolic Syndrome
Brief Title: The Effects of Hesperidin on Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6780
Record Dates: First submitted 2018-10-11; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Hesperidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hesperidin (Active Comparator)
  Interventions: Dietary Supplement: hesperidin
- control (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: hesperidin — 500 mg hesperidin as two capsuls
  Arms: hesperidin
Other: control — no supplementation
  Arms: control

SUMMARY:
To study the effects of Hesperidin supplement in patients with metabolic syndrome, 50 patients will be randomly allocated to control group or 2 capsules Hesperidin for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, metabolic factors will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* having 3 of 5 of high blood sugar, hypertension, high TG, high waist circumference, low HDL

Exclusion Criteria:

* pregnancy or lactation
* A history of Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* Following program to lose weight in recent 3 mo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome: Number of participants with treated metabolic syndrome | 12 weeks
  number of participants with treated metabolic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Yari Z, Movahedian M, Imani H, Alavian SM, Hedayati M, Hekmatdoost A. The effect of hesperidin supplementation on metabolic profiles in patients with metabolic syndrome: a randomized, double-blind, placebo-controlled clinical trial. Eur J Nutr. 2020 Sep;59(6):2569-2577. doi: 10.1007/s00394-019-02105-2. Epub 2019 Dec 16. PMID 31844967